CLINICAL TRIAL: NCT04328792
Title: Prediction Model Based on Deep Learning of CP-EBUS Multimodal Image in the Diagnosis of Benign and Malignant Lymph Nodes
Brief Title: Prediction Model of CP-EBUS in the Diagnosis of Lymph Nodes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director,Department of Respiratory Endoscopy ,Shanghai Chest Hospital, Shanghai Chest Hospital
Other Study IDs: SHCHE201906
Record Dates: First submitted 2019-12-02; First posted 2020-03-31 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Lymph Node Disease
Keywords: EBUS-TBNA; Intrathoracic lymph node; Multimodal image; Deep learning; Prediction model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospectively validation group: Two diagnosis methods will be used in the prospective validation section, one is traditional qualitative and quantitative method, the other is artificial intelligence prediction model based on videos to compare the diagnostic efficacy.

SUMMARY:
Endobronchial ultrasound (EBUS) multimodal image including grey scale, blood flow doppler and elastography, can be used as non-invasive diagnosis and supplement the pathological result, which has important clinical application value. In this study, EBUS multimodal image database of 1000 inthoracic benign and malignant lymph nodes (LNs) will be constructed to train deep learning neural networks, which can automatically select representative images and diagnose LNs. Investigators will establish an artificial intelligence prediction model based on deep learning of intrathoracic LNs, and verify the model in other 300 LNs.

DETAILED DESCRIPTION:
Intrathoracic LNs enlargement has a wide range of diseases, among which intrathoracic LNs metastasis of lung cancer is the most common malignant disease. Benign lesions, including inflammation, tuberculosis and sarcoidosis, also need to be differentiated for targeted treatment.

EBUS multimodal image including grey scale, blood flow doppler and elastography, can be used as non-invasive diagnosis and supplement the pathological result, which has important clinical application value. This study includes two parts: retrospectively construction of EBUS artificial intelligence prediction model and multi-center prospectively validation of the prediction model. A total of 1300 LNs will be enrolled in the study.

During the retention of videos, target LNs and peripheral vessels are examined using ultrasound hosts (EU-ME2, Olympus or Hi-vision Avius, Hitachi) equipped with elastography and doppler functions and ultrasound bronchoscopy (BF-UC260FW, Olympus or EB1970UK, Pentax). Multimodal image data of target LNs are collected.

Investigators will construct artificial intelligence prediction model based on deep learning using images from 1000 LNs firstly, and verify the model in other 300 LNs. This model will be compared with traditional qualitative and quantitative evaluation methods to verify the diagnostic efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Chest CT shows enlarged intrathoracic LNs (short diameter > 1 cm) or PET / CT shows patients with increased FDG uptake (SUV ≧ 2.0) in intrathoracic LNs;
2. Operating physician considered EBUS-TBNA should be performed on LNs for diagnosis or preoperative staging of lung cancer;
3. Patients agree to undergo EBUS-TBNA, sign informed consent, and have no contraindications.

Exclusion Criteria:

- Patients having other situations that are not suitable for EBUS-TBNA.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with enlarged intrathoracic LNs that need to be diagnosed by EBUS-TBNA are enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy of EBUS multimodal artificial intelligence prediction model based on videos | 6 months post-procedure
  Diagnostic efficacy includes sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy.

SECONDARY OUTCOMES:
Diagnostic efficacy of traditional qualitative and quantitative methods | 6 months post-procedure
  Diagnostic efficacy includes sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy.
Diagnostic efficacy of multimodal deep learning model based on images | 6 months post-procedure
  Diagnostic efficacy includes sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy.
Comparion of prediction model based on deeping learning with traditional qualitative and quantitative methods | 6 months post-procedure
  Diagnostic efficacy includes sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, PhD, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Investigators may release the database after the study, but no decision has been made yet.

REFERENCES:
- [Background] Steinfort DP, Conron M, Tsui A, Pasricha SR, Renwick WE, Antippa P, Irving LB. Endobronchial ultrasound-guided transbronchial needle aspiration for the evaluation of suspected lymphoma. J Thorac Oncol. 2010 Jun;5(6):804-9. doi: 10.1097/jto.0b013e3181d873be. PMID 20521347
- [Background] Sun J, Teng J, Yang H, Li Z, Zhang J, Zhao H, Garfield DH, Han B. Endobronchial ultrasound-guided transbronchial needle aspiration in diagnosing intrathoracic tuberculosis. Ann Thorac Surg. 2013 Dec;96(6):2021-7. doi: 10.1016/j.athoracsur.2013.07.005. Epub 2013 Sep 12. PMID 24035300
- [Background] Fujiwara T, Yasufuku K, Nakajima T, Chiyo M, Yoshida S, Suzuki M, Shibuya K, Hiroshima K, Nakatani Y, Yoshino I. The utility of sonographic features during endobronchial ultrasound-guided transbronchial needle aspiration for lymph node staging in patients with lung cancer: a standard endobronchial ultrasound image classification system. Chest. 2010 Sep;138(3):641-7. doi: 10.1378/chest.09-2006. Epub 2010 Apr 9. PMID 20382710
- [Background] Nakajima T, Anayama T, Shingyoji M, Kimura H, Yoshino I, Yasufuku K. Vascular image patterns of lymph nodes for the prediction of metastatic disease during EBUS-TBNA for mediastinal staging of lung cancer. J Thorac Oncol. 2012 Jun;7(6):1009-14. doi: 10.1097/JTO.0b013e31824cbafa. PMID 22525556
- [Background] Wang L, Wu W, Hu Y, Teng J, Zhong R, Han B, Sun J. Sonographic Features of Endobronchial Ultrasonography Predict Intrathoracic Lymph Node Metastasis in Lung Cancer Patients. Ann Thorac Surg. 2015 Oct;100(4):1203-9. doi: 10.1016/j.athoracsur.2015.04.143. Epub 2015 Jul 28. PMID 26228606
- [Background] Izumo T, Sasada S, Chavez C, Matsumoto Y, Tsuchida T. Endobronchial ultrasound elastography in the diagnosis of mediastinal and hilar lymph nodes. Jpn J Clin Oncol. 2014 Oct;44(10):956-62. doi: 10.1093/jjco/hyu105. Epub 2014 Aug 13. PMID 25121724
- [Background] Saftoiu A, Vilmann P, Gorunescu F, Janssen J, Hocke M, Larsen M, Iglesias-Garcia J, Arcidiacono P, Will U, Giovannini M, Dietrich C, Havre R, Gheorghe C, McKay C, Gheonea DI, Ciurea T; European EUS Elastography Multicentric Study Group. Accuracy of endoscopic ultrasound elastography used for differential diagnosis of focal pancreatic masses: a multicenter study. Endoscopy. 2011 Jul;43(7):596-603. doi: 10.1055/s-0030-1256314. Epub 2011 Mar 24. PMID 21437851
- [Background] Gulshan V, Peng L, Coram M, Stumpe MC, Wu D, Narayanaswamy A, Venugopalan S, Widner K, Madams T, Cuadros J, Kim R, Raman R, Nelson PC, Mega JL, Webster DR. Development and Validation of a Deep Learning Algorithm for Detection of Diabetic Retinopathy in Retinal Fundus Photographs. JAMA. 2016 Dec 13;316(22):2402-2410. doi: 10.1001/jama.2016.17216. PMID 27898976